CLINICAL TRIAL: NCT04832490
Title: Early Results of ULD CT-scan for Extremity in Emergency Room
Brief Title: ULD-E (Ultra Low Dose Extremities)
Acronym: ULD E
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Principal Investigator, Ahmed Larbi, hospital practitioner, Centre Hospitalier Universitaire de Nīmes
Other Study IDs: Local 2018/AL
Record Dates: First submitted 2021-03-23; First posted 2021-04-05 (Actual); Last update posted 2021-04-05 (Actual); Status verified 2021-04

CONDITIONS: Wounds and Injuries, Hands; Wounds and Injuries, Wrists; Wounds and Injuries, Feet; Wounds and Injuries, Ankles
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
extremity trauma is a frequent reason for emergency room visits. There is an increase in the use of CT scanners in extremity trauma, due to a greater sensitivity of detection than X-rays, particularly for "occult fractures" and for the organization of treatment, particularly surgical treatment. As the number of CT scans increases, the reduction of the delivered dose has become a subject of interest.

Among the many methods used, the use of iterative reconstruction has enabled a substantial reduction in the delivered dose without compromising image quality: low-dose and ultra-low-dose protocols (effective dose equivalent to the effective dose of the Diagnostic Reference Levels of radiographs from the same region of interest) have been developped, but have not yet been evaluated in extremity trauma.

The subject of our feasibility study is to evaluate the diagnostic performance of ultra-low dose CT compared to radiographs in patients consulting for extremity trauma in the emergency room.

The recent implementation in our department of a scanner dedicated to low-dose explorations as well as the optimization of protocols has allowed the realization of ultra-low-dose scans since June 2017.

DETAILED DESCRIPTION:
The study included all consecutive adult patients who consulted for trauma to the extremities, i.e. hands and wrists, feet and ankles, in the emergency department between February and August 2018. Patients included had undergone digital radiography and ULD-CT for a diagnosis of trauma during weekdays, during working hours (9am-6pm), excluding weekends and holidays. Patients with severe polytrauma requiring a whole body CT scan and patients for whom digital radiography was not the first imaging modality performed were not included in the study.

ULD-CT images were acquired using a Somatom Definition AS+ CT-scan (Siemens Healthineers). Acquisition parameters were as follows: beam collimation of 64×0.6 mm; field of view of 500 mm; pitch factor of 0.85; rotation time of 1.0 s. The tube voltage was fixed at 80 kVp, and the tube current was set at 12 mAs for hands and wrists and at 15 mAs for feet and ankles. Both the automatic adjustment of tube voltage (CARE kV) and the automatic tube current modulation (CARE Dose4D) were disabled. The images were reconstructed in transverse plane of 1-mm thickness and 0.7mm overlapping, and raw data were reconstructed using the level 4 of the SAFIRE® (Sinogram Affirmed Iterative Reconstruction) algorithm. The reconstruction kernels used were "moderately smooth" (I30f) for soft tissue exploration and "strongly sharp" (I70f) for bone exploration for all locations.

Imaging interpretation Image analysis and interpretation were performed retrospectively in a blinded manner by two radiologists, a junior reader with a 3-year experience (TA, reader 1) and a senior reader with a 11-year experience (FS, reader 2). The two radiologists separately analyzed all radiographs after image anonymization and randomization of the reading rank. To limit interpretation biases, a period of 4 weeks was observed before interpretation of the ULD-CT images. They were analyzed separately by the two same radiologists, in the same blinded manner than radiographs, also after randomization of the reading rank. The images were visualized on GE Healthcare Centricity Picture Archiving and Communication System (PACS); all ULD-CT images were read in multiplanar 3-mm reconstructed slices.

ELIGIBILITY:
Inclusion Criteria:

* Major patients consulting in the emergency room of the Nîmes University Hospital during working hours
* Extremity Trauma: Hands/wrists Feet/ankles

Exclusion Criteria:

* opposition to trial participation
* Minor patients
* Polytraumatized patient with body scanner considered

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study included all consecutive adult patients consulting for trauma of the extremities, i.e. hands and wrists and feet and ankles, at the emergency department. Patients included had underwent both digital radiography and ULD-CT for trauma diagnosis during week days, within working hours (9am-6pm), excluding week-ends and public holidays. Patients with severe polytraumas requiring a whole body-scan and patients for whom digital radiography was not the first imaging modality performed were not included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2018-08-01 (Actual); Study Completion 2018-08-01 (Actual)

PRIMARY OUTCOMES:
presence or not of fracture | 1 year
  number of fractures detected after consensus interpretation of the two readers

CONTACTS AND LOCATIONS:
Locations (1):
- Takieddine ADDALA, Nîmes, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Addala TE, Greffier J, Hamard A, Snene F, Bobbia X, Bastide S, Belaouni A, de Forges H, Larbi A, de la Coussaye JE, Beregi JP, Claret PG, Frandon J. Early results of ultra-low-dose CT-scan for extremity traumas in emergency room. Quant Imaging Med Surg. 2022 Aug;12(8):4248-4258. doi: 10.21037/qims-21-848. PMID 35919065